CLINICAL TRIAL: NCT00276718
Title: Germ Cell Tumour Study II
Brief Title: Etoposide, Carboplatin, and Bleomycin in Treating Young Patients Undergoing Surgery For Malignant Germ Cell Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454749; CCLG-GC-1989-01; EU-20583
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-02

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Ovarian Cancer
Keywords: childhood malignant ovarian germ cell tumor; childhood malignant testicular germ cell tumor; childhood central nervous system germ cell tumor; childhood extragonadal germ cell tumor; childhood teratoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Ovarian Neoplasms; Ovarian Germ Cell Cancer; Testicular Neoplasms; Teratoma | interventions — Bleomycin; Carboplatin; Etoposide

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: carboplatin
Drug: etoposide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as etoposide, carboplatin, and bleomycin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving chemotherapy drugs before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving combination chemotherapy after surgery may kill any tumor cells that remain.

PURPOSE: This clinical trial is studying how well giving etoposide, carboplatin, and bleomycin works in treating young patients undergoing surgery for malignant germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects of etoposide, carboplatin, and bleomycin in young patients with malignant germ cell tumors.

OUTLINE: Patients are assigned to one of two treatment arms based on their tumor type (testicular vs ovarian, uterine, vaginal, sacrococcygeal, retroperitoneal, or thoracic).

* Group 1 (testicular tumors): Patients undergo radical orchiectomy. Patients with stage I tumors and alpha-fetoprotein (AFP) decreasing at the expected rate receive no further treatment unless there is a subsequent rise in the AFP or a clinical recurrence. Patients with stage II-IV tumors receive etoposide IV over 1 hour on days 1-3, carboplatin IV over 1 hour on day 2, and bleomycin IV over 15 minutes on day 3. Treatment repeats every 21- 28 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Residual teratoma may be removed, if indicated, after completion of chemotherapy.
* Group 2 (ovarian, uterine, vaginal, sacrococcygeal, retroperitoneal, or thoracic germ cell tumors): Patients undergo surgical removal or biopsy of the tumor. Patients then receive etoposide, carboplatin, and bleomycin as above. Patients may then undergo further surgery at the discretion of the principal investigator.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignant germ cell tumors at all stages

  * Testicular tumors

    * Stage I - Confined to testes
    * Stage II - Confined to testes and retroperitoneal/abdominal lymph nodes
    * Stage III - Supradiaphragmatic nodal disease (mediastinal and/or supraclavicular)
    * Stage IV - Extralymphatic spread (liver, lung, bone, brain, skin, etc.)
  * Ovarian, uterine, vaginal, and sacrococcygeal tumors

    * Stage I - Confined to ovary/uterus/vagina/pre- and postsacral area
    * Stage II - Spread limited to the pelvis
    * Stage III - Spread limited to the abdomen (excluding liver)
    * Stage IV - Spread to liver or beyond the abdominal cavity
  * Abdominal, retroperitoneal, and thoracic primary tumors

    * Stage I - Confined to site of origin and resectable
    * Stage II - Local spread
    * Stage III - Extensive spread confined to one side of the diaphragm (excluding the liver)
    * Stage IV - Tumor spread to the liver, to both sides of the diaphragm, and/or to bones, bone marrow, brain, etc.
  * Intracranial germ cell tumor cases allowed even if an alternative protocol is being followed

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 1989-04

CONTACTS AND LOCATIONS:
Overall Officials: A. Oakhill, MD, Study Chair — Bristol Royal Hospital for Children; Michael Sokal — Nottingham City Hospital; P. Gornall, MD — Birmingham Children's Hospital
Locations (22):
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales